CLINICAL TRIAL: NCT02444195
Title: Self-Administered Guided Imagery in the Perioperative Period to Reduce Postoperative Distress in Gynecologic Oncology Patients: A Randomized Control Trial
Brief Title: Guided Imagery in the Perioperative Period in Gynecologic Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Brandy Michaels, Gynecologic Oncology Fellow, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00095520
Record Dates: First submitted 2015-05-07; First posted 2015-05-14 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Uterine Cervical Neoplasms; Uterine Neoplasms; Ovarian Neoplasms; Urogenital Neoplasms; Fallopian Tube Neoplasms
Keywords: gynecologic cancer; guided imagery; postoperative distress; perioperative distress
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Ovarian Neoplasms; Urogenital Neoplasms; Fallopian Tube Neoplasms | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guided Imagery (Experimental): Guided Imagery With Audio Media
  Interventions: Behavioral: Guided Imagery With Audio Media
- Routine Postoperative Care (No Intervention): Subjects will receive routine pre-operative, intra-operative, post-operative, chemotherapy, and radiation care as dictated by pathologic diagnosis.

INTERVENTIONS:
Behavioral: Guided Imagery With Audio Media — Subjects assigned to the experimental arm will be asked to participate in meditation daily using the audio media provided for the 7 days prior to surgery, in the preoperative holding area, for the 7 days following surgery, and are encouraged to engage in affirmations module use at least weekly in the 6-8 week postoperative period.
  Arms: Guided Imagery

SUMMARY:
The purpose of this study is to evaluate the effectiveness of self-administered perioperative guided imagery to reduce perioperative distress in gynecologic oncology patients undergoing surgical management for a presumed cancer diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgical management for a suspected diagnosis of Gynecologic Malignancy (Endometrial, Ovarian, Vulvar, Vaginal, Primary Peritoneal, Fallopian Tube)
* Age 18 or greater
* Receiving care at University of Michigan Comprehensive Cancer Center Gynecologic Oncology Clinic or at St. Joseph Mercy Hospital, Alexander Cancer Care Center
* Able to understand and read English
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients must have working telephone, mobile or land line

Exclusion Criteria:

* Severe hearing impairment that limits the ability to use audio-based guided imagery modules
* Current documented alcohol abuse or illicit drug substance abuse
* Planned outpatient surgery
* Patients currently participating in a meditation practice for more than 1 hour per week prior to preoperative visit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Level of distress in the immediate postoperative period, measured by the numeric rating scale/ National Comprehensive Cancer Network (NCCN) Distress Thermometer screening instrument. | postoperative day 1
Level of distress in the delayed postoperative period, measured by the numeric rating scale/ National Comprehensive Cancer Network (NCCN) Distress Thermometer screening instrument. | 6-8 week postoperative exam

SECONDARY OUTCOMES:
Level of distress, measured by questionnaire using the Hospital Anxiety and Depression Scale-total (HADS-T). | postoperative day 1 and 6-8 week postoperative exam
Level of anxiety and depressions, measured by questionnaire using the Hospital Anxiety and Depression Scale subscale for anxiety (HADS-A) and depression (HADS-D). | postoperative day 1 and 6-8 week postoperative exam
Level of pain, measured by a 7-item questionnaire using a Likert numerical rating scale for pain | postoperative day 1 and 6-8 week postoperative exam
Perioperative analgesic use, measured by patient-completed usage log and hospital medical record. | postoperative day 1 and 6-8 week postoperative exam
Patient satisfaction regarding in hospital perioperative care, measured by a questionnaire adapted from the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) survey. | postoperative day 1 and 6-8 week postoperative exam
Effect of perioperative guided imagery on health care compliance, measured by the General Adherence Scale (GAS) survey. | 6-8 week postoperative visit
Effect of perioperative guided imagery on health care related locus of control, measured by the Multidimensional Health Locus of Control-form A (MHLC-A) questionnaire. | postoperative day 1 and 6-8 week postoperative exam
The effect of perioperative guided imagery on hope, measured by the Adult Hope Scale (AHS) questionnaire. | postoperative day 1 and 6-8 week postoperative exam

CONTACTS AND LOCATIONS:
Overall Officials: Brandy Michaels, MD, Principal Investigator — University of Michigan; J. Rebecca Liu, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No